CLINICAL TRIAL: NCT01284881
Title: Self-Reported vs Objective Measured Compliance With Oral Appliance Therapy for Obstructive Sleep Apnea Hypopnea Syndrome
Brief Title: Self-Reported Versus Objective Measured Compliance With Oral Appliance Therapy for Obstructive Sleep Apnea Hypopnea Syndrome
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Ethisch Comité UZ Antwerpen, Ethical Comité Antwerp, University Hospital, Antwerp
Other Study IDs: EC 10/42/284
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: OSAHS
Keywords: MRA; compliance; OSAHS
MeSH Terms: conditions — Sleep Apnea, Obstructive; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OSAHS
  Interventions: Device: MRA

INTERVENTIONS:
Device: MRA — daily wear overnight

SUMMARY:
Oral appliances, such as Mandibular Repositioning Appliances (MRA), have emerged as a treatment option for sleep-disordered breathing (SDB).

The purpose of this study is to compare active measurement of MRA compliance with patient's self-report.

DETAILED DESCRIPTION:
Background Oral appliances, such as Mandibular Repositioning Appliances (MRA), have emerged as a conservative treatment option for sleep-disordered breathing (SDB).

Up to this date, no objective method is available to measure compliance during oral appliance treatment for SDB.

As with CPAP in the early years, the sleep apnea community nowadays has a strong interest in the objective measurement of oral appliance use and adherence. Subjective measures and self-report commonly result in overestimation of compliance.

Methods We will perform a 12-week clinical trial comparing active/objective measurement of compliance with subjective self-reported usage.

We will enroll 50 patients with an established diagnosis of SDB that received treatment with a titratable, duobloc MRA (RespiDent Butterfly® MRA, RespiDent, Nijlen, Belgium).

Active microsensors (TheraMon®,Handelsagentur Gschladt, Hargelsberg, Oostenrijk) are provided by the Handelsagentr Gschladt (Hargelsberg, Oostenrijk) without any costs. The sampling interval of the recording will be done at a rate of 1 measurement per 15 minutes (every 900 seconds). Using this sample interval, the capacity of the active microsensor allows for data acquisition during a 100 day period.

The microsensors are intercalated into the MRA devices by the dental technician.

Participants receive explanation to the purpose of the study, in the fact that the investigators want to study temperature fluctuations during the night in the oral cavity. As a result, the subjects are unaware that their MRA use and compliance is being measured.

A first follow-up appointment is scheduled after the first 4 weeks. A second and final follow-up visit is scheduled again 12 weeks after the start of the study.

During each follow-up visit patients are asked to fill out a questionnaire containing questions about MRA wear during the last 4 or 8 weeks (mean hours/night, mean nights/week), respectively. The objective measurement of MRA wear time (total hours of wear time and the mean hours of wear per night over the respective period) will be based on the assumption that the MRA has been worn when the chip records a temperature intraorally.

This study design will provide a 12-week evaluation of all patients (n=50).

Perspective and Hypothesis The removable nature of an oral appliance warrants an objective assessment of the effective use and compliance with overnight MRA treatment for SDB.

We hypothesize that objective compliance might turn out to be significantly lower compared to the subjectively reported compliance.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of sleep-disordered breathing
* started treatment with oral appliances, such as mandibular repositioning appliances

Exclusion Criteria:

* dental exclusion criteria for MRA
* medical contra-indications for MRA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: OSAHS
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Belgium

REFERENCES:
- [Derived] Dieltjens M, Verbruggen AE, Braem MJ, Wouters K, Verbraecken JA, De Backer WA, Hamans E, Van de Heyning PH, Vanderveken OM. Determinants of Objective Compliance During Oral Appliance Therapy in Patients With Sleep-Disordered Breathing: A Prospective Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2015 Oct;141(10):894-900. doi: 10.1001/jamaoto.2015.1756. PMID 26402736
- [Derived] Dieltjens M, Braem MJ, Vroegop AVMT, Wouters K, Verbraecken JA, De Backer WA, Van de Heyning PH, Vanderveken OM. Objectively measured vs self-reported compliance during oral appliance therapy for sleep-disordered breathing. Chest. 2013 Nov;144(5):1495-1502. doi: 10.1378/chest.13-0613. PMID 23928873